CLINICAL TRIAL: NCT03682484
Title: A Phase 1 Combined Single and Multiple Ascending Oral Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MA-0211 in Healthy Adult Subjects Including a Food Effect Cohort
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MA-0211 in Healthy Adult Subjects Including a Food Effect Cohort
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0367-CL-0001
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; MA-0211; Single Ascending Dose; Healthy Volunteer; Multiple Ascending Dose; Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MA-0211 Single Ascending Dose (fasting conditions) (Experimental): Successive cohorts of 8 participants (1-7 cohorts) will be started on a fixed single dose of MA-0211 or matching Placebo under fasting conditions. The first two participants will receive either MA-0211 or matching placebo. If no safety issues are observed in the first 24 hours in the first two participants, then the remaining six participants will be dosed.
  Interventions: Drug: MA-0211
- Placebo Single Ascending Dose (fasting conditions) (Placebo Comparator): Successive cohorts of 8 participants (1-7 cohorts) will be started on a fixed single dose of MA-0211 or matching Placebo under fasting conditions. The first two participants will receive either MA-0211 or matching placebo. If no safety issues are observed in the first 24 hours in the first two participants, then the remaining six participants will be dosed.
  Interventions: Drug: Placebo
- MA-0211 Single Ascending Dose (food effect) (Experimental): A single cohort of 8 participants will be started on a fixed single dose of MA-0211, within 30 minutes after the start and 5 minutes after the completion of an US Food and Drug Administration (FDA) high fat breakfast.
  Interventions: Drug: MA-0211
- MA-0211 Multiple Ascending Dose (Experimental): Successive cohorts of 12 participants (1-3 cohorts) will receive oral doses of MA-0211 or matching Placebo for 14 days.
  Interventions: Drug: MA-0211
- Placebo Multiple Ascending Dose (Placebo Comparator): Successive cohorts of 12 participants (1-3 cohorts) will receive oral doses of MA-0211 or matching Placebo for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MA-0211 — oral
  Other Names: ASP0367
  Arms: MA-0211 Multiple Ascending Dose; MA-0211 Single Ascending Dose (fasting conditions); MA-0211 Single Ascending Dose (food effect)
Drug: Placebo — oral
  Arms: Placebo Multiple Ascending Dose; Placebo Single Ascending Dose (fasting conditions)

SUMMARY:
This first-in-human (FiH) study consists of 2 parts: single ascending dose (SAD) with evaluation of food effect (Part 1) and multiple ascending dose (MAD) (Part 2).

The primary purpose of this study is to evaluate the safety and tolerability of single ascending oral doses in Part 1 (SAD Including Evaluation of Food Effect) and multiple ascending oral doses in Part 2 (MAD) of MA-0211 in healthy adult participants.

This study will also evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of single ascending and multiple ascending oral doses of MA-0211 in healthy adult participants. In addition, this study will evaluate the effect of a single oral dose of MA-0211 on the QT interval using Fridericia's Correction (QTcF); determine the effect of food on the PK of a single oral dose of MA-0211 as well as evaluate the effect of multiple oral doses of MA-0211 on the QTcF.

DETAILED DESCRIPTION:
After a screening period of up to 29 days prior to study drug administration, eligible participants will be residential for a single period of 6 days/5 nights in Part 1 and 19 days/18 nights in Part 2 . Participants will be admitted to the clinical unit on day 2.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) range of 18.5 to 32.0 kg/m2, inclusive, and weighs at least 50 kg at screening.
* Female subject must either:

  * Be of nonchildbearing potential: Postmenopausal (defined as at least 1 year without any menses for which there is no other obvious pathological or physiological cause) prior to screening, or documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy)
  * Or, if of childbearing potential, agree not to try to become pregnant during the study and for 28 days after the final study drug administration, and have a negative blood/urine pregnancy test at screening and day -2, and if heterosexually active, agree to consistently use 1 form of highly effective birth control starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* A sexually active male subject with female partner(s) who are of childbearing potential is eligible if:

  * Agree to use a male condom starting at screening and continue throughout study treatment and for 90 days after the final study drug administration. If the male subject has not had a vasectomy or is not sterile as defined below the subject's female partner(s) is utilizing 1 form of highly effective birth control starting at screening and continue throughout study treatment and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period, and for 90 days after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 28 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present clinical study, defined as signing the informed consent form until completion of the last study visit.

Exclusion Criteria:

* Subject participated in any clinical study or has been treated with any investigational drugs within 28 days prior to screening.
* Subject has any condition which makes the subject unsuitable for clinical study participation.
* Female subject who has been pregnant within 6 months prior to screening assessment or breast feeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to MA-0211, or any components of the formulation used.
* Subject has had previous exposure with MA-0211.
* Subject has any of the liver function tests (aspartate aminotransferase [AST], alanine amino-transferase [ALT], alkaline phosphatase [ALP], gamma-glutamyl transferase [GGT] and total bilirubin [TBL]) above the upper limit of normal at day -2. In such a case, the assessment may be repeated once.
* Subject has total creatine kinase greater than 1.5 times the upper limit of normal or troponin I above the upper limit of normal at day -2.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to study drug administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, psychiatric, dermatologic, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to (day -2).
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, ECG and protocol-defined clinical safety laboratory tests at screening or day 2.
* Subject has a mean heart rate < 45 or > 90 beats per minute; mean Systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg at day -2 (vital signs measurements taken in triplicate after subject has been resting in supine position for 5 minutes; heart rate will be measured automatically). If the mean heart rate, SBP or DBP exceeds the limits above, 1 additional triplicate can be taken (day -2).
* Subject has a mean QT interval using Fridericia's correction (QTcF) > 430ms (for males) and >450ms (for females) at day 2 or if the subject has any family history of long QT syndrome (LQTS). If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken (day -2).
* Subject has used any prescribed or nonprescribed drugs (including vitamins, calcium and iron supplements, natural and herbal remedies [e.g., St. John's Wort]) in the 2 weeks (or 5 elimination half-lives, whichever is longer) prior to study drug administration, except for occasional use of acetaminophen (up to 2 g/day [prn]). In addition, subject has used any peroxisome proliferator-activated receptor (PPAR) ligands such as fibrates and thiazolidinediones in the 4 weeks prior to day -2.
* Subject has smoked or has used tobacco-containing products and nicotine or nicotine containing products in the past 6 months prior to screening.
* Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/ substance abuse within the past 2 years prior to screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor) or the subject tests positive for alcohol or drugs of abuse at screening or day -2 (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates).
* Subject has used any drugs of abuse within 3 months prior to day -2.
* Subject has used any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 month prior to day -2.
* Subject has had significant blood loss, donated 1 unit (500 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day -2.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg) and hepatitis B core antibodies (anti-HBc), hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies (anti-HCV) or antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 at screening.
* Subject anticipates an inability to abstain from caffeine-, xanthine- or grapefruit/Seville orange containing products from at least 24 hours (longer for grapefruit/Seville orange containing products: 72 hours) before screening, and from at least 24 hours (longer for grapefruit/Seville orange containing products: 72 hours) before admission to the clinical unit on day -2 up to and including the End of Study Visit (ESV).
* Subject is an employee of the Astellas Group or Clinical Research Organization (CRO).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by nature, frequency, and severity of Adverse Events (AEs) | Up to day 26
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Number of participants with vital sign abnormalities and /or adverse events (AEs) | Up to day 26
  Number of participants with potentially clinically significant vital sign values.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to day 26
  Number of participants with potentially clinically significant laboratory values.
Safety assessed by routine 12- lead electrocardiogram (ECG) | Up to day 26
  The overall conclusion of the routine ECG will be recorded as normal, abnormal not clinically significant, or abnormal clinically significant.
Safety assessed by continuous 12- lead electrocardiogram (ECG) | Up to day 15
  The overall conclusion of the continuous ECG will be recorded as normal or abnormal, with a comment added if abnormal.
Safety assessed by Real-time cardiac monitoring (telemetry) (Part 1) | Day 1
  Number of participants with potentially clinically significant telemetry abnormalities.

SECONDARY OUTCOMES:
Part 1: Pharmacokinetics (PK) of MA-0211 in plasma: area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf) | Up to day 6
  AUCinf will be derived from the PK plasma samples collected.
Part 1: PK of MA-0211 in plasma: area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast) | Up to day 6
  AUClast will be derived from the PK plasma samples collected.
Part 1: PK of MA-0211 in plasma: percentage of AUCinf due to extrapolation from time of the last measurable concentration to time infinity (AUCinf(%extrap)) | Up to day 6
  AUCinf(%extrap) will be derived from the PK plasma samples collected.
Part 1: PK of MA-0211 in plasma: maximum concentration (Cmax) | Up to day 6
  Cmax will be derived from the PK plasma samples collected.
Part 2 (Only First Dose and Last Dose): PK of MA-0211 in plasma: maximum concentration (Cmax) | Up to day 19
  Cmax will be derived from the PK plasma samples collected.
Part 1: PK of MA-0211 in plasma: time prior to the time corresponding to the first measurable (nonzero) concentration (tlag) | Up to day 6
  tlag will be derived from the PK plasma samples collected.
Part 2 (Only First Dose): PK of MA-0211 in plasma: time prior to the time corresponding to the first measurable (nonzero) concentration (tlag) | Up to day 19
  tlag will be derived from the PK plasma samples collected.
Part 1: PK of MA-0211 in plasma: time of maximum concentration (tmax) | Up to day 6
  tmax will be derived from the PK plasma samples collected.
Part 2 (Only First Dose and Last Dose): PK of MA-0211 in plasma: time of maximum concentration (tmax) | Up to day 19
  tmax will be derived from the PK plasma samples collected.
Part 1: PK of MA-0211 in plasma: apparent total systemic clearance after extravascular dosing (CL/F) | Up to day 6
  CL/F will be derived from the PK plasma samples collected.
Part 2 (Only Last Dose): PK of MA-0211 in plasma: apparent total systemic clearance after extravascular dosing (CL/F) | Up to day 19
  CL/F will be derived from the PK plasma samples collected.
Part 1: PK of MA-0211 in plasma: terminal elimination half-life (t ½) | Up to day 6
  t ½ will be derived from the PK plasma samples collected.
Part 2 (Only Last Dose): PK of MA-0211 in plasma: terminal elimination half-life (t ½) | Up to day 19
  t ½ will be derived from the PK plasma samples collected.
Part 1: PK of MA-0211 in plasma: apparent volume of distribution during the terminal elimination phase after extravascular dosing (Vz/F) | Up to day 6
  Vz/F will be derived from the PK plasma samples collected.
Part 2 (Only Last Dose): PK of MA-0211 in plasma: apparent volume of distribution during the terminal elimination phase after extravascular dosing (Vz/F) | Up to day 19
  Vz/F will be derived from the PK plasma samples collected.
Part 2: PK of MA-0211 in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to day 15
  Ctrough will be derived from the PK plasma samples collected.
Part 2 (Only First Dose): PK of MA-0211 in plasma: area under the concentration-time curve from the time of dosing to 24 hours postdose (AUC24) | Up to day 19
  AUC24 will be derived from the PK plasma samples collected.
Part 2 (Only Last Dose): PK of MA-0211 in plasma Area under the curve over a dosing interval (AUCtau) | Up to day 19
  AUCtau will be derived from the PK plasma samples collected.
Part 2 (Only Last Dose): PK of MA-0211 in plasma: peak-trough ratio (PTR) | Up to day 19
  PTR will be derived from the PK plasma samples collected.
Part 2 (Only Last Dose): PK of MA-0211 in plasma: accumulation ratio calculated using the area under the concentration-time curve (Rac(AUC)) | Up to day 19
  Rac(AUC) will be derived from the PK plasma samples collected.
Part 1: Pharmacodynamic (PD) of MA-0211: Twelve peroxisome proliferator-activated receptor (PPAR) delta target genes expression levels | Up to day 2
  To assess the PD of MA-0211 in Part 1.
Part 2: (Only First Dose and Last Dose) PD of MA-0211: Twelve peroxisome proliferator-activated receptor (PPAR) delta target genes expression levels | Up to day 15
  To assess the PD of MA-0211 in Part 2.
Part 2: (Only First Dose and Last Dose) PD of MA-0211: Serum myostatin | Up to day 15
  To assess the PD of MA-0211 in Part 2.
Part 2: (Only First Dose and Last Dose) PD of MA-0211: follistatin levels | Up to day 15
  To assess the PD of MA-0211 in Part 2.
Part 2: PD of MA-0211: Plasma acyl-carnitine levels | Up to day 15
  To assess the PD of MA-0211 in Part 2.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Parexel - Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.